CLINICAL TRIAL: NCT05622123
Title: The Effects of Faecal Microbiota Transplantation on Beta Cell Preservation in Patients With Newly Diagnosed Type 1 Diabetes
Brief Title: BetaFIT Study: Beta Cell Imaging After Faecal mIcrobiota Transplantation
Acronym: BetaFIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL81554.091.22
Record Dates: First submitted 2022-11-08; First posted 2022-11-18 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2022-11

CONDITIONS: Type 1 Diabetes
Keywords: Faecal microbiota transplantation; GLP-1 receptor; exendin; beta cell mass; beta cell function; imaging; microbiome
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — (Nle14,Lys40(Ahx-NODAGA-68Ga)NH2)exendin-4

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with type 1 diabetes who have completed the ENCAPSULATE-DM1 or FMT preserve-DM1 trial (Experimental): PET/CT imaging after injection with 68Ga-NODAGA-exendin-4 to quantify beta cell mass
  Interventions: Drug: 68Ga-NODAGA-Exendin-4

INTERVENTIONS:
Drug: 68Ga-NODAGA-Exendin-4 — PET/CT imaging after injection with 68Ga-NODAGA-exendin-4

SUMMARY:
The main goal is to investigate whether beta cell mass is correlated to beta cell function after autologous faecal microbial transplantation (FMT) in patients with newly diagnosed type 1 diabetes

DETAILED DESCRIPTION:
The incidence of Type 1 Diabetes Mellitus (T1D) has tripled in the last thirty years, and T1D is associated with a lifelong increase of considerable morbidity and mortality compared to healthy subjects. As the increased T1D incidence is primarily observed in subjects who are not genetically predisposed, environmental factors including altered diet, antibiotic use as well as mode of birth have been suggested to play a role, and these factors have invariably been linked to changes in the gut microbiome. Indeed, an altered composition of the faecal microbiota composition was observed in adolescent T1D patients. A previous study by de Groot et al. (2021) showed that faecal microbiota transplantation stops the decline in endogenous insulin production in newly diagnosed type 1 diabetes patients. However, it is unknown whether this is due to an increase in beta cell mass, or increased function of the remaining beta cells.

In this study, the investigators aim to investigate whether beta cell mass (quantified by 68Ga-NODAGA-exendin-4 PET/CT imaging) is correlated to beta cell function after autologous faecal microbial transplantation in patients with newly diagnosed type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Previously participated in ENCAPSULATE-DM1 or FMT preserve-DM1 trial
* Type 1 diabetes with the diagnosis being made in the last 4.5 years
* Presence of at least one autoantibody associated with type 1 diabetes (anti-GAD-65, anti-IA2, islet cell antibodies, insulin autoantibodies)
* Age ≥ 18 years
* BMI 18-30 kg/m2
* Insulin use

Exclusion Criteria:

* Inability to provide written informed consent
* Other medication use than insulin
* Smoking
* Evidence of compromised immunity
* Presence of a second autoimmune disease (other than type 1 diabetes); e.g. celiac disease, hyper- or hypothyroidism, inflammatory bowel disease. Vitiligo is allowed.
* Pregnancy or the wish to become pregnant within 1 month after the study
* Breastfeeding
* Liver disease defined as aspartate aminotransferase or alanine aminotransferase level of more than three times the upper limit of normal range
* Renal disease defined as MDRD < 40 ml/min/1.73 m²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between residual beta cell mass and function | 1 year
  The correlation between residual beta cell mass measured with 68Ga-NODAGA-Exendin-4 PET/CT imaging at 12 ±1 months and beta cell function derived in the ENCAPSULATE-DM1 or FMT preserve-DM1

SECONDARY OUTCOMES:
Correlation with other parameters | 1 year
  Beta cell mass will be related to parameters derived in the ENCAPSULATE-DM1 or FMT preserve-DM1 study (e.g. immunity status, insulin sensitivity)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gotthardt, MD, Prof., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands